CLINICAL TRIAL: NCT02380482
Title: Myocardial Dysfunction at Early Phase of Traumatic Brain Injury : Evaluation by Two Dimensional and Speckle Tracking Transthoracic Echocardiography
Acronym: Echo-TC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Echo-TC
Record Dates: First submitted 2015-02-23; First posted 2015-03-05 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic brain injury; Myocardial dysfunction; Transthoracic echocardiography; Speckle tracking
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traumatic brain injury (Other): Two dimensional and speckle tracking transthoracic echocardiography in traumatic brain injured patients
  * Glasgow score < or = 9 or
  * Glasgow score between 9 and 13 (included) and Following Traumatic Coma Data Bank Tomographic Damages:
  diffuse injuries type III or IV or mass lesion over 25ml and/or neurosurgical injuries
  Interventions: Other: Transthoracic echocardiography on TBI patients
- Controls (Other): Two dimensional and speckle tracking transthoracic echocardiography in control patients paired with traumatic brain injured patient on age, BMI and sex with the following criteria:
  * Intubated and mechanically ventilated
  * Undergoing urgent non severe surgery
  Interventions: Other: Transthoracic echocardiography on control patients

INTERVENTIONS:
Other: Transthoracic echocardiography on TBI patients — Two Dimensional and speckle trackingTransthoracic echocardiography on TBI patients within 24 hours of trauma
  Arms: Traumatic brain injury
Other: Transthoracic echocardiography on control patients — Two Dimensional and speckle trackingTransthoracic echocardiography on control patients while intubated-ventilated
  Arms: Controls

SUMMARY:
Traumatic brain injury (TBI) is a frequent pathology leading to major morbidity and mortality in young people. Cerebral flood flow maintenance is a major goal directed therapy to improve the prognosis of the patient. Due to cerebral-myocardial interaction, a myocardial dysfunction might occur at the early phase of the traumatic brain injury. This myocardial dysfunction could be partly responsible for a decrease in cerebral blood flow. In such case, improving myocardial dysfunction may help to increase cerebral blood flow and improve patient prognosis. In clinical practice the easiest and non invasive way to explore myocardial dysfunction is with transthoracic echocardiography. The objective of this trial is to investigate myocardial dysfunction at the early phase of traumatic brain injury, compared with a controlled group without TBI.

ELIGIBILITY:
TBI patients

Inclusion Criteria:

* Isolated and non opened traumatic brain injury
* 18 - 65 years old
* Intubated and mechanically ventilated
* Glasgow score < or = 9 or
* Glasgow score between 9 and 13 (included) and Following Traumatic Coma Data Bank Tomographic Damages diffuse injuries type III or IV or mass lesion over 25ml and/or neurosurgical injuries
* Medical insurance

Exclusion Criteria:

* Treated major cardiovascular risks factors
* cardiovascular past medical history (acute cardiovascular event)
* Cardio thoracic surgery
* Brain dead status
* Inotrope drugs
* Severe polytraumatism
* Acute haemorrhage
* Non echogenic patient
* High level athlete
* Incapacitated person by law and pregnant women
* Discovery during echocardiography of underlying cardiomyopathy
* Urgent neurosurgery required

Control patients

Inclusion Criteria:

* Isolated and non opened traumatic brain injury
* 18 - 65 years old
* Intubated and mechanically ventilated
* Paired with TBI patient on age, BMI and sex
* Undergoing urgent non severe surgery
* Medical insurance

Exclusion Criteria:

* Traumatic brain injury
* Treated major cardiovascular risks factors
* cardiovascular past medical history (acute cardiovascular event)
* Cardio thoracic surgery
* Inotrope and vasopressive drugs
* Circulatory failure
* Non echogenic patient
* High level athlete
* Incapacitated person by law and pregnant women
* Discovery during echocardiography of underlying cardiomyopathy
* Urgent neurosurgery required

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-12; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
left ventricular ejection fraction | within the first 24 hours after injury

SECONDARY OUTCOMES:
Strain evaluation by speckle tracking (in percentage of systolic duration) | within the first 24 hours after injury
Systolic strain rate by speckle tracking (in second) | within the first 24 hours after injury
Diastolic strain rate by speckle tracking (in second) | within the first 24 hours after injury
Systolic rotational velocity by speckle tracking (in degree by second) | within the first 24 hours after injury
Diastolic rotational velocity by speckle tracking (in degree by second) | within the first 24 hours after injury
Systolic twisting velocity by speckle tracking (in degree by second) | within the first 24 hours after injury
Diastolic untwisting velocity by speckle tracking (in degree by second) | within the first 24 hours after injury
Myocardial wall thickness (in millimeter) | within the first 24 hours after injury
  2D transthoracic echography
left ventricular diastolic function (cm/sec) | within the first 24 hours after injury
  2D transthoracic echography
Cardiac index | within the first 24 hours after injury
  2D transthoracic echography
tissue doppler imaging (cm/sec) | within the first 24 hours after injury
  2D transthoracic echography
right ventricular diastolic function | within the first 24 hours after injury
  2D transthoracic echography
right ventricular systolic function | within the first 24 hours after injury
  2D transthoracic echography

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital, Grenoble, France

REFERENCES:
- [Background] Bahloul M, Chaari AN, Kallel H, Khabir A, Ayadi A, Charfeddine H, Hergafi L, Chaari AD, Chelly HE, Ben Hamida C, Rekik N, Bouaziz M. Neurogenic pulmonary edema due to traumatic brain injury: evidence of cardiac dysfunction. Am J Crit Care. 2006 Sep;15(5):462-70. PMID 16926367
- [Background] Eagle KA, Berger PB, Calkins H, Chaitman BR, Ewy GA, Fleischmann KE, Fleisher LA, Froehlich JB, Gusberg RJ, Leppo JA, Ryan T, Schlant RC, Winters WL Jr, Gibbons RJ, Antman EM, Alpert JS, Faxon DP, Fuster V, Gregoratos G, Jacobs AK, Hiratzka LF, Russell RO, Smith SC Jr; American College of Cardiology; American Heart Association. ACC/AHA guideline update for perioperative cardiovascular evaluation for noncardiac surgery--executive summary: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee to Update the 1996 Guidelines on Perioperative Cardiovascular Evaluation for Noncardiac Surgery). J Am Coll Cardiol. 2002 Feb 6;39(3):542-53. doi: 10.1016/s0735-1097(01)01788-0. No abstract available. PMID 11823097
- [Background] Lang RM, Bierig M, Devereux RB, Flachskampf FA, Foster E, Pellikka PA, Picard MH, Roman MJ, Seward J, Shanewise JS, Solomon SD, Spencer KT, Sutton MS, Stewart WJ; Chamber Quantification Writing Group; American Society of Echocardiography's Guidelines and Standards Committee; European Association of Echocardiography. Recommendations for chamber quantification: a report from the American Society of Echocardiography's Guidelines and Standards Committee and the Chamber Quantification Writing Group, developed in conjunction with the European Association of Echocardiography, a branch of the European Society of Cardiology. J Am Soc Echocardiogr. 2005 Dec;18(12):1440-63. doi: 10.1016/j.echo.2005.10.005. No abstract available. PMID 16376782
- [Background] Mor-Avi V, Lang RM, Badano LP, Belohlavek M, Cardim NM, Derumeaux G, Galderisi M, Marwick T, Nagueh SF, Sengupta PP, Sicari R, Smiseth OA, Smulevitz B, Takeuchi M, Thomas JD, Vannan M, Voigt JU, Zamorano JL. Current and evolving echocardiographic techniques for the quantitative evaluation of cardiac mechanics: ASE/EAE consensus statement on methodology and indications endorsed by the Japanese Society of Echocardiography. J Am Soc Echocardiogr. 2011 Mar;24(3):277-313. doi: 10.1016/j.echo.2011.01.015. PMID 21338865
- [Background] Moussouttas M, Lai EW, Khoury J, Huynh TT, Dombrowski K, Pacak K. Determinants of central sympathetic activation in spontaneous primary subarachnoid hemorrhage. Neurocrit Care. 2012 Jun;16(3):381-8. doi: 10.1007/s12028-012-9673-5. PMID 22311230
- [Background] Prathep S, Sharma D, Hallman M, Joffe A, Krishnamoorthy V, Mackensen GB, Vavilala MS. Preliminary report on cardiac dysfunction after isolated traumatic brain injury. Crit Care Med. 2014 Jan;42(1):142-7. doi: 10.1097/CCM.0b013e318298a890. PMID 23963125
- [Background] Rosenthal G, Hemphill JC 3rd, Sorani M, Martin C, Morabito D, Obrist WD, Manley GT. Brain tissue oxygen tension is more indicative of oxygen diffusion than oxygen delivery and metabolism in patients with traumatic brain injury. Crit Care Med. 2008 Jun;36(6):1917-24. doi: 10.1097/CCM.0b013e3181743d77. PMID 18496376
- [Background] Schrader H, Hall C, Zwetnow NN. Effects of prolonged supratentorial mass expansion on regional blood flow and cardiovascular parameters during the Cushing response. Acta Neurol Scand. 1985 Sep;72(3):283-94. doi: 10.1111/j.1600-0404.1985.tb00872.x. PMID 4061050
- [Background] Shanlin RJ, Sole MJ, Rahimifar M, Tator CH, Factor SM. Increased intracranial pressure elicits hypertension, increased sympathetic activity, electrocardiographic abnormalities and myocardial damage in rats. J Am Coll Cardiol. 1988 Sep;12(3):727-36. doi: 10.1016/s0735-1097(88)80065-2. PMID 3403832
- [Background] Shivalkar B, Van Loon J, Wieland W, Tjandra-Maga TB, Borgers M, Plets C, Flameng W. Variable effects of explosive or gradual increase of intracranial pressure on myocardial structure and function. Circulation. 1993 Jan;87(1):230-9. doi: 10.1161/01.cir.87.1.230. PMID 8419012
- [Background] Song HS, Back JH, Jin DK, Chung PW, Moon HS, Suh BC, Kim YB, Kim BM, Woo HY, Lee YT, Park KY. Cardiac troponin T elevation after stroke: relationships between elevated serum troponin T, stroke location, and prognosis. J Clin Neurol. 2008 Jun;4(2):75-83. doi: 10.3988/jcn.2008.4.2.75. Epub 2008 Jun 20. PMID 19513307
- [Background] Sosin DM, Sniezek JE, Waxweiler RJ. Trends in death associated with traumatic brain injury, 1979 through 1992. Success and failure. JAMA. 1995 Jun 14;273(22):1778-80. PMID 7769773
- [Derived] Cuisinier A, Maufrais C, Payen JF, Nottin S, Walther G, Bouzat P. Myocardial function at the early phase of traumatic brain injury: a prospective controlled study. Scand J Trauma Resusc Emerg Med. 2016 Oct 28;24(1):129. doi: 10.1186/s13049-016-0323-3. PMID 27793208